CLINICAL TRIAL: NCT07372586
Title: Integration of a Behavioral Health Collaborative Care Model Into an ICU Recovery Clinic
Brief Title: Behavioral Health Collaborative Care Model in an ICU Recovery Clinic
Acronym: BeColM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Health Resources and Services Administration (HRSA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Rita Bakhru, Associate Professor-Faculty, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00145295
Record Dates: First submitted 2026-01-12; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: PICS; Anxiety; Depression - Major Depressive Disorder; Post-Traumatic Stress; PTSD; Critical Illness Recovery; Critical Illness; Collaborative Care; Behavioral Health Concerns
Keywords: critical illness; post-ICU; PICS; anxiety; depression; PTSD; collaborative care model; behavioral health
MeSH Terms: conditions — Anxiety Disorders; Stress Disorders, Post-Traumatic; Critical Illness; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Attention Control
- Interventional (Experimental)
  Interventions: Behavioral: Behavioral Health Collaborative Care Model

INTERVENTIONS:
Behavioral: Behavioral Health Collaborative Care Model — behavioral health collaborative care model in ICU recovery patients and families
  Arms: Interventional

SUMMARY:
Survivors of critical illness are at high risk for mental health issues such as anxiety, depression, and PTSD. This single-site, randomized controlled trial at the Medical University of South Carolina will enroll 150 patients to compare outcomes between a behavioral health Collaborative Care Model (BH CoCM) and usual care (attention control). The intervention includes digital tools (Neuroflow), behavioral health coaching, and psychiatric support.

DETAILED DESCRIPTION:
Patients seen in the MUSC ICU Recovery Clinic will be approached for consent for enrollment. Patients that consent will be randomized to an attention control group or an intervention group.

The intervention group receive BH CoCM. They will have access to NeuroFlow platform, which has been specifically designed to support delivery of a BH CoCM. They will utilize Neuroflow for 6 months. They will undergo assessments for anxiety, depression, post-traumatic stress. A behavioral manager will monitor their needs and provide behavioral health coaching and psychiatric support as needed.

The attention control group will undergo assessments for anxiety, depression, post-traumatic stress.

Investigators will look at changes over six months in intervention group compared to attention control group for patients in terms of symptoms of depression, anxiety, post-traumatic stress. Investigators will also look at adherence, BH CoCM implementation metrics, type and amount of guided content accessed in NeuroFlow. Investigators will perform qualitative surveys to understand better what patients thought about the intervention and ways in which it could be improved.

ELIGIBILITY:
Inclusion Criteria:

- Attendance at the MUSC ICU Recovery Clinic within 180 days of discharge from the hospital

Exclusion Criteria:

* ICU Admission was due to a primary addiction diagnosis (eg alcohol withdrawal or delirium tremens requiring ICU care)
* Serious Mental Illness such as Schizophrenia, psychotic disorder, acute mania
* Late Stage Dementia or Cognitive Impairment
* Limited English or Spanish Proficiency
* Lack of regular access to a computer, tablet or mobile device with internet access

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-01-13 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Depression | Enrollment to 6 months
  Changes over six months in intervention group compared to attention control group for patients in terms of symptoms of depression (PHQ-9: Patient Health Questionnaire-9).
Anxiety | enrollment to six months
  Changes over six months in intervention group compared to attention control group for patients in terms of symptoms of anxiety (GAD-7: Generalized Anxiety Disorder 7)
Post-Traumatic Stress | enrollment to six months
  Changes over six months in intervention group compared to attention control group for patients in terms of symptoms of post-traumatic stress (PCL-5:Patient Health Questionnaire-9).

CONTACTS AND LOCATIONS:
Overall Officials: Rita Bakhru, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No